CLINICAL TRIAL: NCT07130305
Title: is There an Effect of Addition of Body Vibration to Intake of Vitamin D on Some Outcomes of Familial Mediterranean Fever
Brief Title: is There an Effect of Adding Body Vibration to Intake of Vitamin D on Some Outcomes of Familial Mediterranean Fever
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-33
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vibration group (Experimental): vibration group OF FMF will contain 20 FMF adolescent girls. who will receive vitamin D and their traditional colchicine doses daily for six months. vibration group will receive also three sessions of 20-min whole body vibration in the week for 6 months
  Interventions: Other: whole body vibration plus usual care
- control group (Active Comparator): control group of Familial mediterranean fever (20 FMF adolescent girls ) will receive vitamin D and their traditional colchicine doses daily for six months.
  Interventions: Other: usual care

INTERVENTIONS:
Other: whole body vibration plus usual care — Familial mediterranean fever (20 FMF adolescent girls ) will be in this vibration group who will receive vitamin D and their traditional colchicine doses daily for six months. vibration group will also receive three sessions of 20-min whole body vibration in the week for 6 months
  Arms: vibration group
Other: usual care — Familial mediterranean fever (20 FMF adolescent girls ) will be in this control group who will receive vitamin D and their traditional colchicine doses daily for six months.
  Arms: control group

SUMMARY:
Familial mediterranean fever (FMF) is common in mediterranean region. this disorder is connected with deterioration in functional performance, fitness of cardiorespiration, muscle strength, and bone mass

DETAILED DESCRIPTION:
Familial mediterranean fever (FMF adolescent girls ) will be collected to be cateogarized to vibration group (vibration group) or control grouping. every group OF FMF will contain 20 FMF adolescent girls. both groups will receive vitamin D and their traditional colchicine doses daily for six months. vibration group will receive three sessions of 20-min whole body vibration in the week for 6 months

ELIGIBILITY:
Inclusion Criteria:

FMF adolecent girls ages 13 -17 years forty patients

Exclusion Criteria:

cardiac problems renal problems liver problems diabetes brain problems

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-01-08 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
bone mineral density | it will be measured after 6 months
  it is a measure for bone density at 2-4 lumbar vertebrae

SECONDARY OUTCOMES:
z score | it will be measured after 6 months
  it is a score for measure for bone mass at 2-4 lumbar vertebrae
vitamin D | it will be measured after 6 months
  it will measured in plasma as serum 25-hydroxyvitamin D
osteoprotegerin | it will be measured after 6 months
  it will measured in plasma
quadriceps torque | it will be measured after 6 months
  it will measured in dominant side
Standing long jump test | it will be measured after 6 months
  it is an indicator for functional performance
Thirty second sit to stand test | it will be measured after 6 months
  it is an indicator for functional performance
Ruffier index | it will be measured after 6 months
  it is an indicator for cardiorespirtory fittness

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Dokki, Egypt